CLINICAL TRIAL: NCT04989699
Title: A Prospective Multicenter, Double-Masked, Randomized, Parallel-Group, Study to Evaluate the Safety, Tolerability, and Efficacy of OTX-TKI (Axitinib Implant) for Intravitreal Use in Subjects With Neovascular Age-Related Macular Degeneration (nAMD)
Brief Title: Study Evaluating the Treatment of OTX-TKI for Subjects With Neovascular Age-related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OTX-TKI-2020-101
Record Dates: First submitted 2021-07-02; First posted 2021-08-04 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Neovascular Age-Related Macular Degeneration
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Intervention Model Description: 3:1
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OTX-TKI (Active Comparator)
  Interventions: Drug: OTX-TKI/Sham
- Aflibercept (Active Comparator)
  Interventions: Drug: Aflibercept/Sham

INTERVENTIONS:
Drug: OTX-TKI/Sham — OTX-TKI is one dose so subsequent visits will be sham to maintain the mask
  Arms: OTX-TKI
Drug: Aflibercept/Sham — Aflibercept administered every 8 weeks
  Other Names: Eylea
  Arms: Aflibercept

SUMMARY:
Evaluate the safety, tolerability, and efficacy of OTX-TKI for intravitreal use in subjects with Neovascular Age-Related Macular Degeneration

DETAILED DESCRIPTION:
Multicenter, double masked, randomized, parallel-group study to evaluate the safety, tolerability, and efficacy of OTX-TKI for intravitreal use in subjects with Neovascular Age-Related Macular Degeneration

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis, within 3 years of screening, of previously treated subfoveal neovascularization (SFNV) secondary to nAMD with leakage involving the fovea, previously treated with documented evidence of an initially favorable clinical response to anti-VEGF therapy (i.e. aflibercept, ranibizumab, brolucizumab, or bevacizumab).
* The macular appearance on OCT is considered to be free of excess intraretinal and/or subretinal fluid as judged by the investigator.
* Must have received at least 3 anti-VEGF injections in the past year.
* Have received the most recent anti-VEGF injection within the past 1-4 weeks prior to screening visit.
* BCVA ETDRS score between 24 and 83 letters (~20/25 to ~20/320 Snellen equivalent)

Exclusion Criteria:

* Have evidence of a scar, fibrosis or atrophy of >50% of the total lesion in the study eye
* Have presence of a disease other than choroidal neovascular membrane (CNVM) due to AMD in the study eye that could affect vision or safety assessments
* Have monocular vision (fellow eye Snellen BCVA is 20/200 or worse

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | Through study completion, an average of 1 year
  Incidence and severity of treatment emergent adverse events

SECONDARY OUTCOMES:
BCVA changes | Through study completion, an average of 1 year
  BCVA Changes from Baseline
Central subfield thickness changes | Through study completion, an average of 1 year
  Central subfield thickness changes from baseline
Rescue Therapy | Through study completion, an average of 1 year
  Proportion of subjects receiving rescue therapy
Absence of Fluid | Through study completion, an average of 1 year
  Proportion of subjects with absence of foveal fluid
Number of injections | Through study completion, an average of 1 year
  Number of injections from baseline

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Ocular Therapeutix, Bakersfield, California
  - Ocular Therapeutix, Oxnard, California
  - Ocular Therapeutix, Altamonte Springs, Florida
  - Ocular Therapeutix, St. Petersburg, Florida
  - Ocular Therapeutix, Reno, Nevada
  - Ocular Therapeutix, The Woodlands, Texas